CLINICAL TRIAL: NCT00330005
Title: A Pilot Study of Psychodynamic Psychotherapy for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFPR-001
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Last update posted 2006-05-25 (Estimated); Status verified 2006-05

CONDITIONS: Bipolar Disorder
Keywords: psychotherapy; bipolar disorder; psychodynamic; psychoeducation; illness management; controlled trial; pilot study
MeSH Terms: conditions — Bipolar Disorder | interventions — Psychotherapy, Group

INTERVENTIONS:
Behavioral: Group Psychotherapy

SUMMARY:
The purpose of this study was to compare a group psychotherapy intervention, the Integrative Outpatient Model, to a convenience control, in adults with bipolar disorder.

DETAILED DESCRIPTION:
The psychotherapy literature suggests that psychological treatments can have a significant impact on the clinical course and outcome for bipolar disorder (Swartz & Frank, 2001). Very few outcome studies have been conducted in group psychotherapy for bipolar disorder, and there are no preliminary studies conducted using the Integrative Outpatient Model, developed specifically for bipolar disorder. Given the lack of preliminary data, a pilot study with a matched-control design is indicated to obtain preliminary data regarding this treatment modality and approach. The IOM is a weekly, long term psychotherapy.

Comparison: Individuals who participate in group psychotherapy will be compared to a control group on mood and symptom ratings, up to 1 year post intervention.

ELIGIBILITY:
Inclusion Criteria:bipolar disorder; functioning level appropriate for outpatient group psychotherapy; willingness to engage in a psychotherapeutic intervention -

Exclusion Criteria: cognitive impairment; prominent psychosis; under 18 years old

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2002-07; Study Completion 2005-01

PRIMARY OUTCOMES:
depression symptoms
manic symptoms
number of days without a bipolar mood episode
global assessment of functioning
clinical global impression for bipolar disorder

CONTACTS AND LOCATIONS:
Overall Officials: Jodi M Gonzalez, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center - Department of Psychiatry, San Antonio, Texas, United States